CLINICAL TRIAL: NCT07199855
Title: Blinatumomab Combined With Venetoclax as Maintenance Therapy After Allo-HSCT in High-risk Ph Negative Acute B-cell Lymphoblastic Leukemia：a Prospective，Single-arm Study
Brief Title: Blinatumomab Combined With Venetoclax as Maintenance Therapy After Allo-HSCT in High-risk Ph Negative Acute B-cell Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xianbo Huang, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250105C
Record Dates: First submitted 2025-09-09; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Adult
Keywords: Philadelphia chromosome-negative;; B-cell Acute Lymphoblastic Leukemia; Blinatumomab; Venetoclax; Allogeneic Hematopoietic Stem Cell Transplantation; maintenance therapy
MeSH Terms: conditions — Burkitt Lymphoma | interventions — venetoclax; Maintenance

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- blinatumomab combined with venetoclax as maintenance therapy (Experimental): blinatumomab combined with venetoclax as maintenance therapy for high-risk Philadelphia chromosome-negative acute B-cell lymphoblastic leukemia (B-ALL) after allogeneic hematopoietic stem cell transplantation
  Interventions: Drug: blinatumomab combined with venetoclax as maintenance therapy

INTERVENTIONS:
Drug: blinatumomab combined with venetoclax as maintenance therapy — blinatumomab combined with venetoclax as maintenance therapy for high-risk Philadelphia chromosome-negative acute B-cell lymphoblastic leukemia (B-ALL) after allogeneic hematopoietic stem cell transplantation

SUMMARY:
This study is a single-center, single-arm, prospective clinical trial evaluating the efficacy and safety of blinatumomab combined with venetoclax as maintenance therapy for high-risk Philadelphia chromosome-negative acute B-cell lymphoblastic leukemia (B-ALL) after allogeneic hematopoietic stem cell transplantation .

DETAILED DESCRIPTION:
This study focuses on high-risk Philadelphia chromosome-negative (Ph-) acute B-cell lymphoblastic leukemia (B-ALL) patients. The primary objective is to evaluate the efficacy of blinatumomab combined with venetoclax as maintenance therapy following allogeneic hematopoietic stem cell transplantation (allo-HSCT) in these patients, while the secondary objective is to assess its safety. The primary endpoint is the 2-year progression-free survival (PFS) rate post-transplantation. Secondary endpoints include the 2-year cumulative relapse rate, 2-year overall survival (OS), incidence of acute graft-versus-host disease (GVHD) within 180 days post-transplant, cumulative incidence of chronic GVHD, graft-versus-host disease-free and relapse-free survival (GRFS), non-relapse mortality (NRM), and the incidence of treatment-emergent adverse events (TEAEs) (defined as occurring from the start of maintenance therapy to 3 months after completion). Safety assessments include the incidence of adverse events and serious adverse events during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Demographics : Patients aged 14-65 years, regardless of gender or race.
* Diagnosis : Confirmed Ph-negative acute B-cell lymphoblastic leukemia (Ph- B-ALL) through bone marrow cytomorphology, cytochemistry, immunophenotyping, chromosomal analysis, and genetic mutation testing, with CD19 surface antigen expression.
* Risk Stratification :

High-risk B-ALL (per NCCN 2024.V2 guidelines) or Standard-risk B-ALL with no pre-transplant remission or Standard-risk B-ALL in first complete remission (CR1) with measurable residual disease (MRD) positivity or Standard-risk B-ALL with ≥CR2 or B-ALL patients receiving reduced-intensity or non-myeloablative conditioning.

* Transplant Eligibility : Scheduled for allogeneic hematopoietic stem cell transplantation (allo-HSCT) with a suitable donor meeting: HLA-identical sibling donor or Unrelated donor (HLA 9-10/10 high-resolution matched) or Haploidentical related donor.
* HCT-CI Score : ≤2 (Hematopoietic Cell Transplantation-Specific Comorbidity Index).
* ECOG Performance Status : ≤2.
* Organ Function :

Serum creatinine ≤1.5×ULN Cardiac ejection fraction ≥50% Baseline SpO₂ >92% Total bilirubin ≤1.5×ULN; ALT/AST ≤2.0×ULN Pulmonary DLCO (hemoglobin-adjusted) ≥40% and FEV1 ≥50%

* Post-Transplant Recovery :

Full donor chimerism Platelet count >50×10⁹/L Absolute neutrophil count >1.0×10⁹/L Hemoglobin >80g/L - Informed Consent : Patient and legal guardian must provide written informed consent, comply with treatment protocols, follow-up visits, and laboratory assessments.

Exclusion Criteria:

* Prior Malignancy : History of malignancy other than acute lymphoblastic leukemia within 5 years, except for adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer post-radical resection, or ductal carcinoma in situ post-resection.
* MRD-Negative B-ALL : Standard-risk B-ALL with MRD-negative status pre-transplant (per NCCN 2024.V2).
* Disease Activity : Relapse of primary disease or CR/MRD positivity (≥0.01%) confirmed by bone marrow re-evaluation within 1 week before maintenance therapy.
* T-Cell Deficiency : Absolute CD3+ T-cell count ≤0.5×10⁹/L prior to maintenance therapy.
* Active GVHD : Concurrent acute/chronic GVHD requiring systemic immunosuppressive treatment.
* Unstable Systemic Diseases : Including but not limited to:
* Unstable angina or cerebrovascular accident/transient ischemic attack (within 3 months)
* Myocardial infarction (within 3 months)
* Congestive heart failure (NYHA Class ≥ III)
* Post-pacemaker implantation with severe arrhythmia requiring medication
* Uncontrolled hepatic/renal/metabolic diseases
* Pulmonary hypertension
* Active Infection : Uncontrolled infections requiring intravenous antibiotics. HIV : Positive human immunodeficiency virus status. Hepatitis : Active HBV/HCV requiring antiviral therapy.
* Psychiatric Conditions : Mental disorders or inability to provide informed consent.
* Substance Abuse : Drug addiction or chronic alcoholism affecting trial evaluation.
* Reproductive Status :

Pregnant/breastfeeding females Fertile patients unwilling to use contraception during treatment and 12 months post-treatment

- Other : Conditions deemed inappropriate by investigators.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
the 2-year progression-free survival (PFS) rate post-transplantation | the 2-year progression-free survival (PFS) rate post-transplantation
  evaluate the 2-year progression-free survival (PFS) rate post-transplantation of blinatumomab combined with venetoclax as maintenance therapy following allogeneic hematopoietic stem cell transplantation (allo-HSCT) in these patients

SECONDARY OUTCOMES:
the 2-year cumulative relapse rate | 2 year after allogeneic hematopoietic stem cell transplantation (allo-HSCT)
2-year overall survival (OS) | 2 year after allogeneic hematopoietic stem cell transplantation (allo-HSCT)

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Tong, Study Director — First Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes